CLINICAL TRIAL: NCT02847260
Title: A 16 Week, Open Label, Multi-centre, Study to Evaluate the Safety, Tolerability and Pharmacodynamic Effects of a Rapid Dose Titration Regimen of Subcutaneous Remodulin® Therapy in Subjects With Pulmonary Arterial Hypertension (PAH)
Brief Title: Safety and Tolerability of Rapid Dose Titration of Subcutaneous Remodulin® Therapy in PAH Subjects (RAPID)
Acronym: RAPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REM-PH-416
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remodulin (Experimental): Remodulin will be initiated, whilst subjects are hospitalized (minimum of 72 hours) and under medical supervision, at approximately 2 ng/kg/min as a continuous SC infusion with dose increments of 1-2 ng/kg/min applied approximately every 12 hours according to clinical response and tolerability. Following discharge, dose rate increments are permitted at 1-2 ng/kg/min with a minimum of 24 hours between each dose up-titration. Once a dose rate of 20 ng/kg/min is achieved, the dose increments can be increased up to 4 ng/kg/min with dose increments separated by at least 24 hours. The aim is to achieve a target dose of 10, 20, and 30 ng/kg/min by the end of weeks 1, 4 and 12, respectively.
  Interventions: Drug: Remodulin

INTERVENTIONS:
Drug: Remodulin — Treatment will be initiated whilst hospitalized at approximately 2.0 ng/kg/min with dose increments of 1- 2 ng/kg/min approximately every 12 hours according to clinical response and tolerability. Following subject discharge, the dose rate is increased by 1-2 ng/kg/min with dose increments separated by at least 24 hours. When a dose rate of 20 ng/kg/min is achieved dose increments can be increased at a rate of up to 4 ng/kg/min with dose increments separated by at least 24 hours depending on tolerability. The aim is to achieve a dose rate of at least 10, 20 and 30 ng/kg/min by the end of weeks 1, 4 and 12, respectively and a dose rate by the end of week 16 that achieves pre-defined treatment goals subject to clinical response and tolerability.
  Other Names: Treprostinil

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a rapid dose titration regimen of subcutaneous Remodulin® therapy in patients with PAH.

DETAILED DESCRIPTION:
This is an open label, single territory, multi-centre study in subjects with pulmonary arterial.

hypertension (PAH). Subjects were treatment naïve or receiving an approved endothelin receptor antagonist (ERA) and / or phosphodiesterase (PDE)-5 inhibitor for at least 60 days prior to screening and maintained on a stable dose for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years of age at screening.
2. The subject weigh a minimum of 40 kg with a body mass index less than 40 kg/m^2 at screening.
3. Sexually active women of childbearing potential must use two different forms of highly effective contraception. Males participating in the study must use a condom during the length of the study, and for at least 64 days after discontinuing study drug.
4. The subject has a diagnosis of symptomatic idiopathic or heritable PAH (IPAH or HPAH).
5. A Baseline 6MWD between 150 and 550 metres is required, in the absence of a concurrent injury, illness (other than PAH or a PAH related condition), or other confounding factors that would effect the subject's exercise capacity.
6. The subject is either treatment naïve or receiving an approved PDE-5 inhibitor and / or an approved ERA for at least 60 days prior to screening and is on a stable dose for 30 days and is willing to remain on a PDE-5 inhibitor and / or an ERA at the same dose for the duration of the 16-week treatment phase.
7. The subject must be optimally treated with conventional pulmonary hypertension therapy (e.g., oral vasodilators, oxygen, digoxin, etc.) with no additions, discontinuations, or dose changes for at least 14 days prior to screening (excluding diuretics and anticoagulant dose adjustments).
8. The subject has undergone right heart catheterisation at screening (or within 8 weeks before screening) and has been documented to have a mean pulmonary artery pressure (PAPm) of greater than or equal to 25 mmHg, a pulmonary capillary wedge pressure (PCWP) of less than or equal to 15 mmHg, and pulmonary vascular resistance (PVR) of more than 3 Wood units.
9. The subject has undergone echocardiography at screening with evidence of clinically normal left systolic and diastolic ventricular function, absence of any clinically significant left sided heart disease (e.g., mitral valve stenosis) and absence of unrepaired congenital heart disease.
10. The subject has a previous ventilation perfusion lung scan and / or high resolution computerised tomography scan of the chest and / or pulmonary angiography that is consistent with the diagnosis of PAH (e.g., low probability of pulmonary embolism; absence of major perfusion defects).
11. The subject has pulmonary function tests done within 9 months of screening with the following:

    * Total lung capacity (TLC) was at least 60% (of predicted value)
    * Forced expiratory volume in one second/forced vital capacity (FEV1/FVC) ratio is at least 50%
12. In the opinion of the Principal Investigator, the subject is able to communicate effectively with study personnel, was considered reliable, willing and likely to be cooperative with protocol requirements.
13. The subject voluntarily gives written informed consent to participate in the study.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject has received epoprostenol, treprostinil, intravenous iloprost, or beraprost within 30 days prior to screening (except if used during acute vasoreactivity testing).
3. The subject has had previous intolerance or significant lack of efficacy to prostacyclin or a prostacyclin analogue that resulted in discontinuation or inability to titrate that therapy effectively.
4. The subject has any disease associated with PH other than idiopathic PAH or heritable PAH or had had an atrial septostomy.
5. The subject is in WHO functional class IV.
6. The subject has a current diagnosis of uncontrolled sleep apnoea as defined by their physician.
7. The subject has liver function tests (aspartate transaminase (AST) or alanine transaminase (ALT)) greater than three times the upper limit of the laboratory reference range and / or an international normalised ratio (INR) greater than 3 units at screening.
8. The subject has a history of active gastro-intestinal ulcer, intracranial haemorrhage, injury or other cause of clinically significant bleeding episode within 6 months before screening, or has any other disease / condition that would either jeopardise the safety of the subject and / or interfere with the interpretation of study assessments in the opinion of the Investigator.
9. The subject has a history of ischemic heart disease including previous myocardial infarction or symptomatic coronary artery disease within 6 months of screening, or history of left sided myocardial disease as evidenced by a PCWP (or Left Ventricular End-Diastolic Pressure (LVEDP)) greater than 15 mmHg or left ventricular ejection fraction (LVEF) less than 40%.
10. The subject has uncontrolled systemic hypertension as evidenced by systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg.
11. The subject has a musculoskeletal disorder (e.g., arthritis affecting the lower limbs, recent hip or knee joint replacement, artificial leg) or any other disease that is likely to limit ambulation, or is connected to a machine that is not portable.
12. The subject has an unstable psychiatric condition or is mentally incapable of understanding the objectives, nature, or consequences of the trial.
13. The subject is receiving an investigational drug, has an investigational device in place or has participated in an investigational drug or device study within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grünig, Principal Investigator — Thoraxklinik am Universitätsklinikum, Heidelberg, Germany; Klose, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany; Rosenkranz, Principal Investigator — Universitätsklinikum Köln, Köln, Germany; Höffken, Principal Investigator — Universitaetsklinikum Dresden, Dresden, Germany; Lange, Principal Investigator — Universitätsklinikum Regensburg, Regensburg, Germany; Wirtz, Principal Investigator — Universitätsklinikum Leipzig, Leipzig, Germany; Neurohr, Principal Investigator — Klinikum Großhadern der LMU, Munich, Germany; Wilkens, Principal Investigator — Universitätsklinikum Klinik, Homburg, Germany; Held, Principal Investigator — Missionsärztliche Klinik, Würzburg, Germany; Krüger, Principal Investigator — Herzzentrum Duisburg, Duisburg, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Remodulin: Remodulin was initiated, whilst subjects were hospitalized, at approximately 2 ng/kg/min as a continuous SC infusion with dose increments of 1-2 ng/kg/min applied approximately every 12 hours according to clinical response and tolerability. Following discharge, dose rate increments were permitted at 1-2 ng/kg/min with a minimum of 24 hours between each dose up-titration. Once a dose rate of 20 ng/kg/min was achieved, the dose increments could be increased up to 4 ng/kg/min, with dose increments separated by at least 24 hours. The aim was to achieve a target dose rate of 10, 20, and 30 ng/kg/min by the end of Weeks 1, 4, and 12, respectively.
Period: Overall Study
Arm/Group | Remodulin
Started | 39
Completed | 32
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Clinical Deterioration | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Remodulin
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 50 [25 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 10
Region of Enrollment [Number; unit: participants]
  Germany | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Completion of the 16 Week Treatment Period.
Description: Successful completion was defined as completion of the 16 week treatment period of the study without experiencing any serious adverse events considered by the investigator to be possibly related to Remodulin.
Time Frame: Baseline to week 16
Measure: Number; unit: participants
Arm/Group | Remodulin
Number analyzed (Participants) | 39
participants | 32

2. Secondary Outcome: Change From Baseline in Six Minute Walk Distance at Week 16.
Description: The purpose of the six minute walk test (6MWT) was to evaluate exercise capacity associated with carrying out activities of daily living. Patients were instructed to walk down a corridor at a comfortable speed as far as they could manage for six minutes, resting whenever they needed. Distance <500 meters suggests considerable exercise limitation; Distance 500 - 800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation.
Time Frame: Baseline to week 16
Population: Two subjects that completed the treatment period did not complete the six minute walk test at week 16. As such, the evaluable data for the six minute walk test at Week 16 was summarized using an N of 30 subjects.
Measure: Median (Full Range); unit: meters
Arm/Group | Remodulin
Number analyzed (Participants) | 30
meters | 11.5 [-62 to 246]

3. Secondary Outcome: Change in Borg Dyspnea Score (Following 6MWT) From Baseline to Week 16
Description: The Borg dyspnea score is a 10 point scale rating the maximum level of dyspnea (difficulty in breathing) experienced during the 6MWT. The Borg dyspnea score was assessed immediately following the 6MWT. Scores range from 0 (for no shortness of breath) to 10 (for the greatest shortness of breath ever experienced).
Time Frame: Baseline to week 16
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Remodulin
Number analyzed (Participants) | 30
units on a scale | 0.0 [-4 to 2]

4. Secondary Outcome: Change in N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) Concentrations From Baseline to Week 16.
Description: The level of this biomarker of the (NT-proBNP) serum concentration was assessed to compare the severity of heart failure at Baseline and Week 16.
Time Frame: Baseline to week 16
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Remodulin
Number analyzed (Participants) | 32
pg/mL | -182.0 [-18396 to 9629]

5. Secondary Outcome: Number of Participants With a Change From Baseline World Health Organization (WHO) Functional Classification at Week 16.
Description: The WHO Functional Class of pulmonary hypertension is a physical activity rating scale as follows: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
Time Frame: Baseline to week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Remodulin
Number analyzed (Participants) | 32
Participants
  II to II | 4
  II to III | 1
  III to II | 8
  III to III | 18
  III to IV | 1

6. Secondary Outcome: Change in Quality of Life (QoL) Assessment: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) From Baseline to Week 16.
Description: The CAMPHOR is a health related quality of life instrument validated for pulmonary hypertension that assesses impairment (symptoms), disability (activities) and quality of life. The questionnaire is divided into three sections; Symptoms (Scores 0-25; high scores indicate more symptoms), Activity (Score 0-30; low score indicates good functioning) and Quality of Life (0-25; high scores indicate poor QoL). The sum of these scores equates to the Total score (0-80). In the CAMPHOR scores, negative change scores indicate improvements.
Time Frame: Baseline to week 16
Population: Scores could not be tabulated for one subject due to missing responses to individual questions
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Remodulin
Number analyzed (Participants) | 31
units on a scale
  CAMPHOR total score | -5.0 [-44 to 13]
  Quality of life | -1.0 [-13 to 7]

7. Secondary Outcome: Change From Baseline to Week 16 in Hemodynamic Parameters: Mean Pulmonary Artery Pressure (PAPm), Mean Right Atrial Pressure (RAPm) and Mean Pulmonary Capillary Wedge Pressure (PCWPm).
Description: Pulmonary hypertension, an increase in pressure in the pulmonary vasculature defined as a mean pulmonary artery pressure (PAPm) greater than 25 mmHg at rest or greater than 30 mmHg with exercise, as measured by Swan-Ganz right heart catheterization. The PAPm, RAPm and PCWPm values and their respective changes from Baseline to Week 16 were measured by SwanGanz right heart catheterization and summarized.
Time Frame: Baseline to week 16
Population: Only 29 of the 32 subjects that completed the 16 week treatment period completed these hemodynamic assessments.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Remodulin
Number analyzed (Participants) | 29
mmHG
  PAPm (mmHg) | -3.2 (10.5)
  RAPm (mmHg) | 0.3 (5.6)
  PCWPm (mmHg) | -0.3 (4.6)

8. Secondary Outcome: Change From Baseline to Week 16 in Hemodynamic Parameters: Cardiac Index (CI) (L/Min/m^2)
Description: Cardiac Index (CI) relates the cardiac output (CO) to body surface area (BSA), thus relating heart performance to the size of the individual. The CI values and their respective changes from Baseline to Week 16 were measured by SwanGanz right heart catheterization and summarized.
Time Frame: Baseline to week 16
Population: Only 29 of the 32 subjects that completed the 16 week treatment period completed these hemodynamic assessments.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Remodulin
Number analyzed (Participants) | 29
L/min/m^2 | 0.4 (0.4)

9. Secondary Outcome: Change From Baseline to Week 16 in HemodynamicParameters: Pulmonary Vascular Resistance Index (PVRI) (mmHg*Min*m^2/L)
Description: Pulmonary Vascular Resistance Index (PVRI) is calculated using Mean Pulmonary Arterial Pressure(PAPm), Pulmonary Capillary Wedge Pressure (PCWP) and Cardiac Index (CI ), to provide information about right ventricular load. The PVRI values and their respective changes from Baseline to Week 16 were measured by SwanGanz right heart catheterization.
Time Frame: Baseline to week 16
Population: Only 29 of the 32 subjects that completed the 16 week treatment period completed these hemodynamic assessments.
Measure: Mean (Standard Deviation); unit: mmHg*min*m^2/L
Arm/Group | Remodulin
Number analyzed (Participants) | 29
mmHg*min*m^2/L | -3.5 (4.5)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 16-week study, including the screening and follow-up phase, as well as 30 days post end of study visit.
Groups:
- Remodulin: Remodulin was initiated, whilst subjects were hospitalized, at approximately 2 ng/kg/min as a continuous SC infusion with dose increments of 1-2 ng/kg/min applied approximately every 12 hours according to clinical response and tolerability. Following discharge, dose rate increments were permitted at 1-2 ng/kg/min with a minimum of 24 hours between each dose up-titration. Once a dose rate of 20 ng/kg/min was achieved, the dose increments could be increased up to 4 ng/kg/min, with dose increments separated by at least 24 hours. The aim was to achieve a target dose of 10, 20, and 30 ng/kg/min by the end of Weeks 1, 4, and 12, respectively.
Arm/Group | Remodulin
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 11/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remodulin (N=39)
Right Ventricular Failure (RVF) (Cardiac disorders) | 3 (3)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2)
Diarrhoea, (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Infusion Site Pain (Skin and subcutaneous tissue disorders) | 2 (2)
Rib Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia, bacterial (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remodulin (N=39)
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 28 (28)
Nausea (Gastrointestinal disorders) | 18 (18)
Vomiting (Gastrointestinal disorders) | 15 (16)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Infusion Site Pain (General disorders) | 36 (37)
Infusion Site Erythema (General disorders) | 10 (10)
Oedema Peripheral (General disorders) | 6 (6)
Infusion Site Haemorrhage (General disorders) | 5 (6)
Fatigue (General disorders) | 3 (3)
Infusion Site Irritation (General disorders) | 4 (4)
Infusion Site Swelling (General disorders) | 4 (4)
Local swelling (General disorders) | 3 (4)
Nasopharyngitis (Infections and infestations) | 6 (8)
Infusion Site Infection (Infections and infestations) | 4 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 9 (9)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 27 (28)
Dizziness (Nervous system disorders) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Flushing (Vascular disorders) | 2 (2)
Injection Site Inflammation (General disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Sleep disorder (Psychiatric disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Infusion site abscess (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed, except as provided below. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.